CLINICAL TRIAL: NCT01577420
Title: Reflexology: An Intervention for Advanced Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gwen Wyatt, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 5R01CA104883-05 (NIH); 5R01CA104883-05 (NIH)
Record Dates: First submitted 2012-04-12; First posted 2012-04-13 (Estimated); Last update posted 2012-04-13 (Estimated); Status verified 2012-04

CONDITIONS: Breast Cancer
Keywords: Reflexology; Breast Cancer; Complementary
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): Reflexology Sessions: One session per week performed by certified reflexologist for four consecutive weeks.
  Interventions: Other: Reflexology Sessions
- Group B (Placebo Comparator): Placebo Sessions: One session per week performed by research aide for four consecutive weeks.
  Interventions: Other: Placebo Sessions
- Group C (No Intervention): Control; no foot sessions

INTERVENTIONS:
Other: Reflexology Sessions — One session per week performed by certified reflexologist for four consecutive weeks.
  Arms: Group A
Other: Placebo Sessions — One session per week performed by research aide for four consecutive weeks.
  Arms: Group B

SUMMARY:
The aim of this study is to test a complementary therapy intervention (reflexology) that will assist in improving quality of life (QOL) for women undergoing chemotherapy for late stage (III or IV) breast cancer within the context of conventional medical care. Quality of life will be assessed via intermediate indicators: 1) physical indicators (greater physical functioning, lower presence of symptoms) 2) emotional indicators (greater spirituality, lower anxiety, and lower depressive symptomology); and the outcome indicator of quality of life.

DETAILED DESCRIPTION:
The goal of this study is to test a complementary therapy intervention that will assist in improving quality of life (QOL) for women undergoing chemotherapy for late stage (III and IV) breast cancer within the context of conventional medical care. This longitudinal randomized clinical trial (RCT) will test a three-group design in which participants will continue to receive conventional care. Two groups of the study will involve a single-blinded four-week protocol: Group A will receive reflexology (a specialized foot therapy) from a certified reflexologist; Group B will receive placebo sessions from a research aide. The control group (Group C) will receive conventional medical care alone. The specific aims are: 1) to determine if women who receive either Groups (A or B) of an experimental protocol (reflexology or placebo) report significantly better QOL outcomes (total and subscales) at 7 weeks, 13 weeks, and longitudinally over time, relative to women receiving conventional care alone (Group C); 2) to determine if women who receive Group A of an experimental protocol (reflexology), report significantly better QOL outcomes (total and subscales) at 7 weeks, 13 weeks, and longitudinally over time, relative to women receiving Group B (placebo; 3) to determine if women who receive either Group A or B of an experimental protocol (reflexology or placebo), report significant differences on Intermediate Indicators (physical and emotional), at 7 weeks, 13 weeks, and longitudinally over time, relative to women receiving conventional care alone; and 4) to determine if the Intermediate Indicators mediate the group effect on the QOL outcomes (total and subscales) at 7 weeks. This has the potential of leading to an enhanced system of care through the integration of conventional and scientifically-based complementary therapies. It also focuses on advanced disease that is currently under investigation in terms of supportive care measures. Finally, this study utilizes an improved design over existing work. It is a RCT with adequate numbers to detect group differences, and could ultimately serve as a model for rigorous investigation of other complementary therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stage III or IV breast cancer, or Stage I or II with Metastasis or Recurrence
* Able to perform basic ADLs
* Free of diagnosis of mental illness on chart
* Able to speak and understand English
* Access to a telephone
* Receiving chemotherapy at intake into the study
* Palliative Prognostic Score of 11 or lower
* Oriented to time, place, and person as determined by nurse recruiter

Exclusion Criteria:

* Receiving investigational new drug chemotherapy
* Receiving hospice care at intake
* Living in nursing home or similar facility
* Bedridden
* Undergoing bone marrow transplant
* Regularly using foot massage
* Regularly using reflexology
* Regularly using pedicure with foot massage

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2005-08; Primary Completion 2010-04 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | Baseline to week 13

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Wyatt, PhD, RN, Principal Investigator — Michigan State University
Locations (12):
- United States (12):
  - Evanston Northwestern, Evanston, Illinois
  - Mt. Clemens, Evanston, Illinois
  - Hurley Medical Center, Flint, Michigan
  - GLCI/McLaren, Flint, Michigan
  - St. Joseph Mercy Oakland Hospital, Grand Rapids, Michigan
  - St. Mary's Health Care Center, Grand Rapids, Michigan
  - Great Lakes Cancer Institute (GLCI) MSU, Lansing, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital-Troy Campus, Troy, Michigan
  - St. John Macomb, Warren, Michigan
  - Josephine Ford Cancer Care, Henry Ford Hospital, West Bloomfield, Michigan

REFERENCES:
- [Background] Sikorskii A, Wyatt G, Victorson D, Faulkner G, Rahbar MH. Methodological issues in trials of complementary and alternative medicine interventions. Nurs Res. 2009 Nov-Dec;58(6):444-51. doi: 10.1097/NNR.0b013e3181bf15fe. PMID 19918155
- [Background] Rahbar MH, Wyatt G, Sikorskii A, Victorson D, Ardjomand-Hessabi M. Coordination and management of multisite complementary and alternative medicine (CAM) therapies: experience from a multisite reflexology intervention trial. Contemp Clin Trials. 2011 Sep;32(5):620-9. doi: 10.1016/j.cct.2011.05.015. Epub 2011 Jun 2. PMID 21664296
- [Background] Wyatt G, Sikorskii A, Rahbar MH, Victorson D, Adams L. Intervention fidelity: aspects of complementary and alternative medicine research. Cancer Nurs. 2010 Sep-Oct;33(5):331-42. doi: 10.1097/NCC.0b013e3181d0b4b7. PMID 20467309
- [Result] Sikorskii A, Wyatt GK, Siddiqi AE, Tamkus D. Recruitment and early retention of women with advanced breast cancer in a complementary and alternative medicine trial. Evid Based Complement Alternat Med. 2011;2011:734517. doi: 10.1093/ecam/nep051. Epub 2011 Feb 14. PMID 19620179